CLINICAL TRIAL: NCT02277548
Title: A Pilot Study at a Single-Institution of Pregabalin in the Management of Mucositis Pain in Patients Undergoing Chemoradiation Therapy to the Head and Neck.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: UPCC 43313
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Oropharyngeal Cancer; Squamous Cell Carcinoma to the Head and Neck
Keywords: chemotherapy; radiation therapy
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lyrica at 300 mg per day (Experimental)
  Interventions: Drug: Lyrica 300 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lyrica 300 mg — Lyrica 300 mg per day
  Arms: Lyrica at 300 mg per day
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the efficacy of pregabalin in the management of mucositis pain in patients receiving radiotherapy to the head and neck. Eligible study subjects will be enrolled among those being treated for oropharyngeal cancer with definitive chemotherapy and radiation therapy (photons) to the head and neck in the Department of Radiation Oncology at the University of Pennsylvania.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated for oropharyngeal cancer with undergoing concurrent chemotherapy and radiation therapy (photons) for a histological diagnosis of squamous cell carcinoma to the head and neck at the University of Pennsylvania
* Age at least 18 years old
* Treatment entails significant risk for symptomatic mucositis likely to require opioid analgesia, as per the discretion of treating physician/NP
* Subjects are capable of giving informed consent

Exclusion Criteria:

* Patients anticipated to receive radiation therapy with Protons
* History of hypersensitivity to pregabalin or gabapentin
* History of seizure or currently taking anti-epileptic medication
* Creatinine clearance of less than 30 mL/min by Cockcroft-Gault estimate
* Has another painful condition requiring chronic use of opioid analgesic, gabapentin, or pregabalin
* History of serious mood disorder or attempted suicide as determined by patients history and physical and by using theDepression Screening
* Subjects with a score of greater than 10 or those answering #5 with scores greater than a "0" will be deemed ineligible to be enrolled on study
* History of angioedema
* New York Heart Association class III or IV heart failure
* Platelets of less than 150 mg/dL or history of thrombocytopenia
* The patient has any uncontrolled intercurrent illness including but not limited to psychiatric illness/social situations that would limit compliance or interfere with their ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin McMenamin, MSN, CRNP, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
Period: Overall Study
Arm/Group | Lyrica at 300 mg Per Day | Placebo
Started | 9 | 11
Completed | 9 | 9
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lyrica at 300 mg Per Day | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (14.1) | 56.3 (10.5) | 56.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Average/Cumulative Opioid Dose
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Lyrica at 300 mg Per Day | Placebo
Number analyzed (Participants) | 9 | 9
mg | 32.65306 (49.74759) | 31.60714 (58.5934)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Lyrica at 300 mg Per Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lyrica at 300 mg Per Day (N=9) | Placebo (N=11)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Elevated creatinine, changed to non-qualifying chemotherapy (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT02277548/Prot_SAP_000.pdf